CLINICAL TRIAL: NCT04844424
Title: An Open-Label, Randomized, Crossover Study to Evaluate the Relative Oral Bioavailability, Pharmacokinetics, and Food Effect After Single Dose (for Part 1, Part 3, Part 4 and Part 5) or Multiple-Dose (for Part 2) Administration of JNJ-70033093 (Milvexian) in Healthy Adult Participants Using Tablet, Capsule and Dispersed Tablet Formulations
Brief Title: A Study of JNJ-70033093 (Milvexian) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108999; 70033093THR1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (44):
- Part 1A: Treatment Sequence ABC (Experimental): Participants will receive a single oral Dose 1 of milvexian as direct compression (DC) tablets under fasting conditions (Treatment A) in Treatment Period 1, followed by a single oral Dose 1 of milvexian as roller compacted (RC) tablets under fasting conditions (Treatment B) in Treatment Period 2 and then a single oral Dose 1 of milvexian Phase 2 oral capsules under fasting conditions (Treatment C) in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1A: Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment C in Treatment Period 2 and then Treatment A in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1A: Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment A in Treatment Period 2 and then Treatment B in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1A: Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1, followed by Treatment C in Treatment Period 2 and then Treatment B in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1A: Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2 and then Treatment C in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1A: Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1 followed by Treatment B in Treatment Period 2 and then Treatment A in Treatment Period 3 on Day 1 of each Treatment Period during Part 1A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence DEF (Experimental): Participants will receive a single oral Dose 1 of milvexian as DC oral tablets under fed conditions (Treatment D) in Treatment Period 1, followed by a single oral Dose 1 of milvexian as RC oral tablets under fed conditions (Treatment E) in Treatment Period 2 and then a single oral Dose 1 of milvexian as Phase 2 oral capsules under fed conditions (Treatment F) in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence EFD (Experimental): Participants will receive Treatment E in Treatment Period 1, followed by Treatment F in Treatment Period 2 and then Treatment D in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence FDE (Experimental): Participants will receive Treatment F in Treatment Period 1, followed by Treatment D in Treatment Period 2 and then Treatment E in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence DFE (Experimental): Participants will receive Treatment D in Treatment Period 1, followed by Treatment F in Treatment Period 2 and then Treatment E in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence EDF (Experimental): Participants will receive Treatment E in Treatment Period 1, followed by Treatment D in Treatment Period 2 and then Treatment F in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 1B: Treatment Sequence FED (Experimental): Participants will receive Treatment F in Treatment Period 1, followed by Treatment E in Treatment Period 2 and then Treatment D in Treatment Period 3 on Day 1 of each Treatment Period during Part 1B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 2A: Treatment Sequence GH (Experimental): Participants will receive twice daily (BID) oral Dose 1 of milvexian DC oral tablets (Treatment G) in Treatment Period 1, followed by BID oral Dose 1 of milvexian Phase 2 oral capsule (Treatment H) in Treatment Period 2 up to Day 5 in each Treatment Period during Part 2A. There will be a wash-out period of more than 5 days between the evening dose of Day 5 of Treatment Period 1 and the morning dose of Day 1 of Treatment Period 2.
  Interventions: Drug: Milvexian
- Part 2A: Treatment Sequence HG (Experimental): Participants will receive Treatment H in Treatment Period 1, followed by Treatment G in Treatment Period 2 up to Day 5 in each Treatment Period during Part 2A. There will be a wash-out period of more than 5 days between the evening dose of Day 5 of Treatment Period 1 and the morning dose of Day 1 of Treatment Period 2.
  Interventions: Drug: Milvexian
- Part 2B: Treatment Sequence IJ (Experimental): Participants will receive BID oral Dose 2 of milvexian DC oral tablet (Treatment I) in Treatment Period 1, followed by BID oral Dose 2 of milvexian Phase 2 oral capsule (Treatment J) in Treatment Period 2 up to Day 5 in each Treatment Period during Part 2B. There will be a wash-out period of more than 5 days between the evening dose of Day 5 of Treatment Period 1 and the morning dose of Day 1 of Treatment Period 2.
  Interventions: Drug: Milvexian
- Part 2B: Treatment Sequence JI (Experimental): Participants will receive Treatment J in Treatment Period 1, followed by Treatment I in Treatment Period 2 up to Day 5 in each Treatment Period during Part 2B. There will be a wash-out period of more than 5 days between the evening dose of Day 5 of Treatment Period 1 and the morning dose of Day 1 of Treatment Period 2.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence KLM (Experimental): Participants will receive single oral Dose 1 of milvexian as oral Tablet 1 under fasting conditions (Treatment K) in Treatment Period 1, followed by single oral Dose 1 of milvexian oral Tablet 2 under fasting conditions (Treatment L) in Treatment Period 2 and then single oral Dose 1 of milvexian as Phase 2 oral capsules under fasting conditions (Treatment M) in Treatment Period 3 on Day 1 in each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence LMK (Experimental): Participants will receive Treatment L in Treatment Period 1, followed by Treatment M in Treatment Period 2 and then Treatment K in Treatment Period 3 on Day 1 of each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence MKL (Experimental): Participants will receive Treatment M in Treatment Period 1, followed by Treatment K in Treatment Period 2 and then Treatment L in Treatment Period 3 on Day 1 in each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence KML (Experimental): Participants will receive Treatment K in Treatment Period 1, followed by Treatment M in Treatment Period 2 and then Treatment L in Treatment Period 3 on Day 1 in each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence LKM (Experimental): Participants will receive Treatment L in Treatment Period 1, followed by Treatment K in Treatment Period 2 and then Treatment M in Treatment Period 3 on Day 1 in each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3A: Treatment Sequence MLK (Experimental): Participants will receive Treatment M in Treatment Period 1, followed by Treatment L in Treatment Period 2 and then Treatment K in Treatment Period 3 on Day 1 in each Treatment Period during Part 3A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence NOP (Experimental): Participants will receive single oral Dose 1 of milvexian oral Tablet 1 under fed conditions (Treatment N) in Treatment Period 1, followed by single oral Dose 1 of milvexian oral Tablet 2 under fed conditions (Treatment O) in Treatment Period 2 and then single oral Dose 1 of milvexian Phase 2 oral capsule under fed conditions (Treatment P) in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence OPN (Experimental): Participants will receive Treatment O in Treatment Period 1, followed by Treatment P in Treatment Period 2 and then Treatment N in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence PNO (Experimental): Participants will receive Treatment P in Treatment Period 1, followed by Treatment N in Treatment Period 2 and then Treatment O in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence NPO (Experimental): Participants will receive Treatment N in Treatment Period 1, followed by Treatment P in Treatment Period 2 and then Treatment O in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence ONP (Experimental): Participants will receive Treatment O in Treatment Period 1, followed by Treatment N in Treatment Period 2 and then Treatment P in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 3B: Treatment Sequence PON (Experimental): Participants will receive Treatment P in Treatment Period 1, followed by Treatment O in Treatment Period 2 and then Treatment N in Treatment Period 3 on Day 1 in each Treatment Period during Part 3B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4 A: Treatment Sequence QRS (Experimental): Participants will receive single oral Dose 1 of milvexian as Phase 3 oral tablets under fasting conditions (Treatment Q) in Treatment Period 1, followed by single oral Dose 1 of milvexian as Phase 3 oral tablets under fed conditions (Treatment R) in Treatment Period 2 and then single oral Dose 1 of milvexian as Phase 3 oral tablets under fed conditions (Treatment S) in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4A: Treatment Sequence RSQ (Experimental): Participants will receive Treatment R in Treatment Period 1, followed by Treatment S in Treatment Period 2 and then Treatment Q in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4A: Treatment Sequence SQR (Experimental): Participants will receive Treatment S in Treatment Period 1, followed by Treatment Q in Treatment Period 2 and then Treatment R in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4A: Treatment Sequence QSR (Experimental): Participants will receive Treatment Q in Treatment Period 1, followed by Treatment S in Treatment Period 2 and then Treatment R in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4A: Treatment Sequence RQS (Experimental): Participants will receive Treatment R in Treatment Period 1, followed by Treatment Q in Treatment Period 2 and then Treatment S in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4A: Treatment Sequence SRQ (Experimental): Participants will receive Treatment S in Treatment Period 1, followed by Treatment R in Treatment Period 2 and then Treatment Q in Treatment Period 3 on Day 1 of each Treatment Period during Part 4A. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4B: Treatment Sequence TU (Experimental): Participants will receive single oral Dose 1 of milvexian as Phase 3 oral tablet under fed conditions (Treatment T) in Treatment Period 1, followed by single oral Dose 2 of milvexian as Phase 3 oral tablet under fed conditions (Treatment U) in Treatment Period 2 on Day 1 of each Treatment Period during Part 4B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 4B: Treatment Sequence UT (Experimental): Participants will receive Treatment U in Treatment Period 1, followed by Treatment T in Treatment Period 2 on Day 1 of each Treatment Period during Part 4B. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Subpart 4A: Treatment Sequence VW (Experimental): All participants of Subpart 4A will undertake a mandatory taste assessment on Day 5 of period 3 or Day 15 before the discharge and will receive milvexian tablet dispersed in water without a sweetener orally via syringe (Treatment V) in Treatment Period 1, followed by milvexian tablet dispersed in water with sucralose sweetener orally via syringe (Treatment W) in Treatment Period 2. Participants will cleanse their palates using 2 rinse of mineral water and one unsalted cracker and wait for a time interval of at least 1-2 hours from start of dosing before the next taste round.
  Interventions: Drug: Milvexian
- Subpart 4A: Treatment Sequence WV (Experimental): All participants of Subpart 4A will undertake a mandatory taste assessment on Day 5 of period 3 or Day 15 before the discharge and will receive Treatment W in Treatment Period 1, followed by Treatment V in Treatment Period 2. Participants will cleanse their palates using 2 rinse of mineral water and one unsalted cracker and wait for a time interval of at least 1-2 hours from start of dosing before the next taste round.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence XYZ (Experimental): Participants will receive a single oral Dose 1 of milvexian as DC whole tablets under fasting conditions (Treatment X) in Treatment Period 1 followed by a single oral Dose 1 of milvexian as DC tablets dispersed in water and then mixed with apple sauce under fasting conditions (Treatment Y) in Treatment Period 2 and then a single oral Dose 1 of milvexian as DC tablets dispersed in water administered through a nasogastric (NG) tube under fasting conditions (Treatment Z) in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence YZX (Experimental): Participants will receive Treatment Y in Treatment Period 1 followed by Treatment Z in Treatment Period 2 and then Treatment X in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence ZXY (Experimental): Participants will receive Treatment Z in Treatment Period 1 followed by Treatment X in Treatment Period 2 and then Treatment Y in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence XZY (Experimental): Participants will receive Treatment X in Treatment Period 1 followed by Treatment Z in Treatment Period 2 and then Treatment Y in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence YXZ (Experimental): Participants will receive Treatment Y in Treatment Period 1 followed by Treatment X in Treatment Period 2 and then Treatment Z in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian
- Part 5: Treatment Sequence ZYX (Experimental): Participants will receive Treatment Z in Treatment Period 1 followed by Treatment Y in Treatment Period 2 and then Treatment X in Treatment Period 3 on Day 1 of each Treatment Period during Part 5. There will be a wash-out period of 5 days between Day 1 of adjacent treatment periods.
  Interventions: Drug: Milvexian

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally or via nasogastric route as tablets or capsules.
  Other Names: JNJ-70033093, BMS-986177

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability and food effect of a single dose of milvexian administered as direct compression (DC) oral tablets and roller compacted (RC) oral tablets compared with milvexian administered as Phase 2 oral capsules (Part 1) and of new concept tablets consisting of a single dose of milvexian administered as oral Tablet 1 and Tablet 2 compared with milvexian administered as Phase 2 oral capsules (Part 3) in healthy participants under fasting and fed conditions; to characterize the pharmacokinetics (PK) of multiple twice daily (BID) doses for 5 days of milvexian administered as DC oral tablets and Phase 2 oral capsules in healthy participants (Part 2) and to assess the effects of dosing time and food timing on the PK of single-dose of milvexian Phase 3 oral tablet formulation in healthy participants (Part 4) and to evaluate the relative bioavailability of a single dose of milvexian administered as oral film-coated DC whole tablets, oral film-coated DC tablets dispersed in water and then mixed with apple sauce, and oral film-coated DC tablets dispersed in water and administered as a suspension using a nasogastric (NG) tube in healthy participants under fasting conditions (Part 5).

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and on Day -1 of Treatment Period 1. If there are abnormalities, the investigator may decide that the abnormalities or deviations from normal are not clinically significant, in which case the participant may be included
* Body mass index (BMI equals to [=] weight/height^2) between 18 and 30 kilograms per meter square (kg/m^2) (inclusive), and body weight not less than 50 kg at screening
* Healthy on the basis of safety laboratory tests performed at screening and on Day -1 of Treatment Period 1. If the results of the safety laboratory tests are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant except as specified in Exclusion Criteria 2. This determination must be recorded in the participant's source documents and initialed by the investigator
* A woman must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and urine pregnancy test on Day 1 of Treatment Period 1
* Before randomization, a woman must be either: a) Not of childbearing potential defined as: postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level greater than (>) 40 international units per liter IU/L or milli-international units per milliliter (mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal replacement therapy (HRT), however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient; permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy; b) Of childbearing potential and; practicing a highly effective method of contraception (failure rate of less than [<] 1 percent [%] per year when used consistently and correctly) for at least 3 months prior to the study entry and; agrees to remain on a highly effective method of contraception throughout the study and for at least 34 days after the last dose of study drug
* During the study, a man who is sexually active with a woman of childbearing potential or with a woman who is pregnant must agree to use a barrier method of contraception (example, condom with spermicidal foam/gel/ film/cream/suppository)

Exclusion Criteria:

* History of any known illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol-specified assessments. This may include but is not limited to any known bleeding or clotting disorder, a history of arterial or venous thrombosis, liver or renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplasm, metabolic disturbances, or poor venous access
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry, or urinalysis at screening or on Day -1 of Treatment Period 1 as determined by the investigator or appropriate designee. Any of the following laboratory results outside of the normal ranges specified below at screening or Day -1 of Treatment Period 1 which must be confirmed by repeat: Hemoglobin or hematocrit less than (<) lower limit of normal; Platelet count < lower limit of normal; activated partial thromboplastin time (aPTT) or prothrombin time (PT) >1.2*upper limit of normal (ULN)
* Use of any agent, including but not limited to non-steroidal anti-inflammatory drugs (NSAIDs), aspirin or other anti-platelet agents, anticoagulants, fish oil capsules, ginkgo or any agent that can potentially increase the risk of bleeding within 14 days prior to the first dose of study drug administration
* History of any clinically significant drug or food allergies (such as anaphylaxis or hepatotoxicity) and known allergy to the study drugs or any of the excipients of the formulation
* History of allergy to or unwillingness to consume any component of the standardized high-fat breakfast menu to be provided in this study
* Woman with history of excessive menstrual bleeding as determined by the investigator or appropriate designee
* Does not tolerate venipuncture

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve of Milvexian from Time Zero to Infinity (AUC [0-Infinity]) | Up to 16 months
  AUC (0-infinity) is defined as area under the plasma concentration-time curve of milvexian from time zero to infinity after administration.
Part 2: Area under the Plasma Concentration-time Curve of Milvexian From Time Zero to Time of Last Quantifiable Concentration (AUC [0-Last]) | Up to 16 months
  AUC (0-last) is defined as area under the plasma concentration-time curve of milvexian from time zero to time of last quantifiable concentration after administration.
Maximum Observed Analyte Concentration (Cmax) of Milvexian | Up to 16 months
  Cmax is defined as maximum observed analyte concentration of milvexian.
Parts 1 and 3: AUC (0-Infinity) of Milvexian (Food effect) | Up to 16 months
  AUC (0-infinity) is defined as area under the plasma concentration-time curve of milvexian from time zero to infinity after administration.
Parts 1 and 3: AUC (0-Last) of Milvexian (Food effect) | Up to 16 months
  AUC (0-last) is defined as area under the plasma concentration-time curve of milvexian from time zero to time of last quantifiable concentration after administration.
Parts 1 and 3: Cmax of Milvexian (Food effect) | Up to 16 months
  Cmax is defined as maximum observed analyte concentration of milvexian.
Actual Sampling Time to Reach the Maximum Observed Analyte Concentration (Tmax) of Milvexian | Up to 16 months
  Tmax is defined as the actual sampling time to reach the maximum observed analyte concentration of milvexian.
Parts 1 and 3: Tmax of Milvexian (Food effect) | Up to 16 months
  Tmax is defined as the actual sampling time to reach the maximum observed analyte concentration of milvexian.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 16 months
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency